CLINICAL TRIAL: NCT02960191
Title: Functional Neuroimaging and Genetic Vulnerability to Suicidal Behavior
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficult
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7887
Record Dates: First submitted 2016-08-30; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Suicidal Behavior
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy volunteers (Other): subject with no current or past personal history of psychiatric disorders and about never having carried out suicide attempt
  Interventions: Device: Magnetic resonance imaging (MRI)
- emotional witness (Other): subject having had a personal history of unipolar or bipolar depressive disorder and who have never done in his life attempted suicide
  Interventions: Device: Magnetic resonance imaging (MRI)
- patient suicide (Other): subject having had a personal history of unipolar or bipolar depressive disorder and having realized in his life at least one suicide attempt
  Interventions: Device: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: Magnetic resonance imaging (MRI)

SUMMARY:
The main objective is to highlight, by functional imaging (MRI) dysfunctional brain regions associated with vulnerability to suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* arm suicidal : Personal history of unipolar depressive disorder or bipolar disorder and having realized in his life at least one suicide attempt
* arm emotional Witnesses : Personal history of unipolar depressive disorder or bipolar disorder and have never done in his life attempted suicide
* arm healthy Witnesses : any current or past personal history of psychiatric disorders of Axis I and have never done in his life attempted suicide

Exclusion Criteria:

* Cons-indications to the use of MRI
* Existence of a past history of head trauma with loss of consciousness or neurological brain disorder or secondary neurological suffering suicidal gesture.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
MRI variations | at day 0
  activation of specific brain areas during the procurement of a test decision

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France